CLINICAL TRIAL: NCT02230618
Title: A Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Post Marketing Surveillance (PMS) Study of Ryzodeg™ (Insulin Degludec/Insulin Aspart) to Evaluate Long Term Safety and Efficacy in Patients With Diabetes Mellitus in Routine Clinical Practice in India
Brief Title: Post Marketing Surveillance (PMS) Study of Ryzodeg™ (Insulin Degludec/Insulin Aspart) in Patients With Diabetes Mellitus in Routine Clinical Practice in India
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN5401-4149; U1111-1157-0615 (Other: World Health Organization (WHO)); ENCEPP/SDPP/6587 (Registry Identifier: EU PASS)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ryzodeg™
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Ryzodeg™ will be prescribed by the physician under normal clinical practice conditions and will be obtained/purchased from the chemist based on physician prescription. No treatment given.

SUMMARY:
This study is conducted in Asia. The aim of this study is to evaluate long term safety and efficacy in patients with diabetes mellitus in routine clinical practice in India.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. (Study-related activities are any procedures that are related to recording of data according to the protocol). The historical data including the data before informed consent obtained (e.g., HbA1c (Glycated Haemoglobin ), FPG (Fasting Plasma Glucose), PPPG (Postprandial Plasma Glucose), severe hypoglycaemia before the start of Ryzodeg™ therapy) can be used for baseline data
* Patients with insulin requiring diabetes mellitus and who are scheduled to start treatment with Ryzodeg™ based on the clinical judgment of their treating physician

Exclusion Criteria:

* Known or suspected allergy to Ryzodeg™ any of the active substances or any of the excipients
* Previous participation in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patients who are or have previously been on Ryzodeg™ therapy
* Patients who are participating in other studies or clinical trials
* Patients who are pregnant, breast feeding or have the intention of becoming pregnant within the following 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes where the treating physician has decided to start Ryzodeg™ according to routine clinical practice will qualify for starting treatment with Ryzodeg™.
Sampling Method: Non-Probability Sample
Enrollment: 1029 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Weeks 0-52

SECONDARY OUTCOMES:
Serious Adverse Events (SAEs) | Weeks 0-52
Serious Adverse Drug Reactions (SADRs) | Weeks 0-52
Adverse Drug Reactions (ADRs) | Weeks 0-52
Severe or Blood glucose (BG) Confirmed hypoglycaemia | Weeks 0-52
Change in HbA1c (glycosylated haemoglobin) | Week 0, week 52
Change in Fasting Plasma Glucose (FPG) | Week 0, week 52
Change in Post Prandial Blood/Plasma Glucose (PPBG/PPPG) | Week 0, week 52
The reason for initiating or intensifying treatment with Ryzodeg™ | Week 0 - week 52

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (27):
- India (27):
  - Novo Nordisk Investigational Site, Guntur, Andhra Pradesh
  - Novo Nordisk Investigational Site, Vijayawada, Andhra Pradesh
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Gandhinagar, Gujarat
  - Novo Nordisk Investigational Site, Ghuma, Gujarat
  - Novo Nordisk Investigational Site, Surat, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mangalore, Karnataka
  - Novo Nordisk Investigational Site, Angamaly, Kerala
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Thrissur, Kerala
  - Novo Nordisk Investigational Site, Trivandrum, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Amritsar, Punjab
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Lucknow, Uttar Pradesh
  - Novo Nordisk Investigational Site, Noida, Uttar Pradesh
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Bilāspur
  - Novo Nordisk Investigational Site, Thriruvananthapuram

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com